CLINICAL TRIAL: NCT02495467
Title: A Randomised, Double-blind, Placebo-controlled, Home Use, Cross-over Clinical Trial of Topically-applied Glyceryl Trinitrate (GTN) for the Treatment of Erectile Dysfunction (ED)
Brief Title: Clinical Trial of Topically-applied Glyceryl Trinitrate (GTN) for the Treatment of Erectile Dysfunction (ED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Futura Medical Developments Ltd. (Industry)
Collaborators: Richmond Pharmacology Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FM53
Record Dates: First submitted 2015-06-29; First posted 2015-07-13 (Estimated); Results first posted 2020-01-29 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-01

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Nitroglycerin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MED Placebo then MED2005 (Experimental): Participants first receive MED Placebo to be used at least 4 times during a 4 week period. Following a 1-week treatment-free cross-over period participants receive MED2005 (0.2% glyceryl trinitrate gel) to be used at least 4 times during a 4 week period. Treatments are provided in single unit dose aluminium tubes packed in boxes of 5. Each tube will contain sufficient gel to apply a pea sized amount (approximately 300 mg).
  Interventions: Drug: Glyceryl trinitrate; Drug: MED Placebo
- MED2005 then MED Placebo (Experimental): Participants first receive MED2005 (0.2% glyceryl trinitrate gel) to be used at least 4 times during a 4 week period. Following a 1-week treatment-free cross-over period participants receive MED Placebo to be used at least 4 times during a 4 week period. Treatments are provided in single unit dose aluminium tubes packed in boxes of 5. Each tube will contain sufficient gel to apply a pea sized amount (approximately 300 mg).
  Interventions: Drug: Glyceryl trinitrate; Drug: MED Placebo

INTERVENTIONS:
Drug: Glyceryl trinitrate — At least 4 applications of MED2005 prior to intercourse over a period of 4 weeks
  Other Names: MED2005
Drug: MED Placebo — At least 4 applications of MED2005 prior to intercourse over a period of 4 weeks
  Other Names: MED2005 Vehicle

SUMMARY:
This study is designed to evaluate the efficacy and safety of MED2005, a topically applied glyceryl trinitrate (GTN) gel administered to the penis of male subjects self-diagnosed with erectile dysfunction (ED) immediately before sexual intercourse.

DETAILED DESCRIPTION:
This randomised, double-blind, placebo-controlled cross-over study is designed to evaluate the efficacy and safety of MED2005, a topically applied glyceryl trinitrate (GTN) gel administered to the penis of male subjects immediately before sexual intercourse. Subjects will be male aged between 18 and 70 years of age self-diagnosed with ED. Treatment requires the topical application of a pea sized volume (approximately 300 mg) of a 0.2% (w/w) gel to deliver a dose of 0.6 mg GTN to the glans of the penis. A total of 192 eligible subjects are planned to be enrolled into the study. Subjects will be screened for eligibility during the screening period (Day -45 to Day -2), provide a history of their ED treatments and those deemed eligible and who have a female consenting partner will participate in a run-in-period and two treatment periods (treatment period 1 and 2). The International Index for Erectile Function (IIEF) question 1 -5 and 15 will be used to determine pre-screening eligibility for the subject online. A score of 25 or less will be acceptable for inclusion to the run-in-period. Screening (visit 1) will be conducted over 1 day or may be divided into more than 1 day if wash-out of prior medications is needed. The screening period is applicable for visit 1 Informed consent will be signed by both partners before a couple can be admitted to the study. There will also be a subject and partner training requirement to ensure that the product is applied in an appropriate manner. After refraining from using other ED treatments for at least a period of a week, in the run-in-period (visit 2), subjects and their female partners will make at least 4 intercourse attempts (with a minimum of 1 attempt per week) during a 4 week (± 1 week) period. The subjects and their partners will be asked to complete questionnaires online to record their experiences after each sexual intercourse attempt and at the end of the run-in period. Subjects who cannot comply with the minimum number of sexual attempts verified by completed Sexual Event Profile (SEP) or exceed 25 on the IIEF question 1 -5 and 15 will be excluded from the study. Scores generated from the run-in period will be used as an established baseline in the planned analyses. The run-in period will be completed prior to randomisation and dosing.

In treatment period 1 (visit 3 and visit 4), subjects will be allocated to receive either placebo or MED2005 (0.6 mg GTN) according to a pre-defined randomisation schedule. After refraining from using other ED treatments for at least a period of a week, subjects and their female partner will be trained in the application of the test article and asked to apply the test article immediately prior to sexual intercourse, and to make at least 4 intercourse attempts during a 4 week (± 1 week) period. The subjects and their partners will be asked to complete questionnaires online to record their experiences after each sexual intercourse attempt, and again at the end of each treatment period. Subjects will be asked to return to the Clinical Pharmacology Unit (CPU) after 4 weeks' (± 1 week) to return used and unused test article from the first treatment period, to enable the clinical staff to check compliance and to assess their health status, including assessment of any Adverse Event (AE). At the end of treatment period 1 (visit 4), tubes will be weighed to ensure subject compliance.

Following a 1 week treatment-free cross-over period, the subjects will enter into treatment period 2.

In treatment period 2 (visit 5 and visit 6), subjects will be issued with the alternative test article, either placebo or MED2005 (0.6 mg GTN) according to the pre-defined randomisation code. Training on the application of the test article will be reinforced / repeated and the subject or their female partner will be asked to apply the test article immediately prior to sexual intercourse on at least 4 separate occasions during a 4-week period. After each intercourse attempt the subjects and their partners will be asked to complete questionnaires online to record their experiences after each sexual intercourse attempt, and again at the end of each treatment period.. Subjects will be asked to return to the CPU after 4 weeks' (± 1 week) time to return used and unused test article from the second treatment period, to enable the clinical staff to check compliance and to assess their health status, including assessment of any AEs. At the end of treatment period 2 (visit 6), tubes will be weighed to ensure subject compliance.

Subjects and their female partners will be followed up at 7 day's ± 2 days (visit 7) after the outpatient visit on week 4 of treatment period 2, as necessary, to follow up any on-going AEs.

ELIGIBILITY:
Inclusion Criteria:

1. Male aged between 18 and 70 years of age inclusive.
2. Confirmed self-diagnosis of ED for more than 3 months.
3. IIEF question 1 -5 and 15 score of 25 or less will be acceptable for inclusion to the run-in period.
4. Subject answers "yes" to the question "At home over the past 3 months, have you experienced at least some growth of your penis in response to: (1) mechanical stimulation, or (2) visual stimulation?"
5. In a continuous heterosexual relationship for at least 6 months prior to screening.
6. Documented written informed consent from both subject and his female partner.
7. Both partners must agree to use one of the acceptable methods of contraception listed below:

   * Occlusive cap (diaphragm or cervical/vault caps).
   * Surgical sterilisation (vasectomy with documentation of azoospermia).
   * The female partner uses oral contraceptives, injectable progesterone or subdermal implants.
   * The female partner uses medically prescribed topically-applied transdermal contraceptive patch.
   * The female partner has undergone documented tubal ligation (female sterilisation).
   * The female partner has undergone documented placement of an Intra Uterine Device (IUD).
8. Both partners are capable of understanding and complying with the requirements of the protocol and must have signed the informed consent form.

Exclusion Criteria:

1. Any significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, haematological, endocrinological, metabolic, neurological, psychiatric, or other disease.
2. Any history of an unstable medical or psychiatric condition or using any medication that, in the opinion of the PI, is likely to affect the subject's ability to complete the study or precludes the subject's participation in the study.
3. Any presence of a symptomatic, active urinary tract infection diagnosed by the PI or delegate at screening.
4. Any presence of chronic indwelling urethral catheterization or penile anatomical abnormalities (e.g. penile fibrosis) that would significantly impair erectile function.
5. Any history of operations for Peyronie's disease.
6. Primary hypoactive sexual desire or any history of hypogonadism
7. Any history of radical prostatectomy.
8. Any history of severe / uncontrolled diabetes.
9. Subjects taking two or more anti-hypertensives for the treatment of blood pressure.
10. Subjects with nursing partners, known pregnant partners or wish to become pregnant during the course of the study.
11. Confirmed positive results from urine drug screen or from the alcohol breath test at screening and on admission (Day -1).
12. Subject has recent (last 12 months) clinical evidence of alcoholism or drug abuse.
13. Subject has a positive screen for hepatitis B consisting of Hepatitis B surface antigen (HBsAG), hepatitis C antibody, and human immunodeficiency virus (HIV).
14. Any clinically significant abnormal laboratory, vital signs or other safety findings at screening or on admission.
15. Subjects unwilling to cease use of vacuum devices, intracavernosal injection, Viagra ® or other therapy for ED.
16. Unwillingness of the subject to agree to make four attempts at sexual intercourse on four separate days during each treatment period.
17. Any history of unresponsiveness to Viagra ® treatment due to lack of efficacy with sexual stimulation after multiple attempts of sexual intercourse, or significant side effects excluding visual disturbances of Viagra ®.
18. Less than 4 attempts at sexual intercourse or high IIEF scores (> 25) during the run-in period.
19. Any known hypersensitivity to any component of the investigational product.
20. Subjects who are illiterate or are unable to understand the language in which the online questionnaires are available.
21. Subject has received any investigational product during the 90 days prior to dosing for this study.
22. Subject or their partner cannot communicate reliably with the Investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2015-05-15 (Actual); Primary Completion 2016-07-30 (Actual); Study Completion 2016-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim J Holland, MSc, Study Director — Futura Medical Developments Ltd.; Jörg Täubel, MD FFPM, Principal Investigator — Richmond Pharmacology Limited
Locations (1):
- Richmond Pharmacology Ltd., Croydon, Surrey, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: First Intervention (4 Weeks)
Arm/Group | MED Placebo Then MED2005 | MED2005 Then MED Placebo
Started | 114 | 118
Completed | 114 | 118 (One subject completed visits in treatment Period 1 but never used treatment)
Not Completed | 0 | 0
Period: Washout (1 Week)
Arm/Group | MED Placebo Then MED2005 | MED2005 Then MED Placebo
Started | 114 | 118
Completed | 112 | 116
Not Completed | 2 | 2
Period: Second Intervention (4 Weeks)
Arm/Group | MED Placebo Then MED2005 | MED2005 Then MED Placebo
Started | 112 | 116
Completed | 112 | 113
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Population: Safety Set. A total of 231 subjects made use of the medication at least once and were included in the safety set.
Groups:
- Total: Total of all reporting groups
Arm/Group | MED Placebo Then MED2005 | MED2005 Then MED Placebo | Total
Number analyzed (Participants) | 114 | 117 | 231
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (13.7) | 43.3 (14.7) | 43.0 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 114 | 117 | 231
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 5 | 4 | 9
  Black or African American | 7 | 10 | 17
  White | 97 | 97 | 194
  Other | 5 | 6 | 11
Erectile Function (EF) domain score of the International Index of Erectile Function (IIEF) [Mean (Standard Deviation); unit: score on a scale] — Erectile Function (EF) domain of the International Index of Erectile Function (IIEF) questionnaire. Measured at the end of a 4 week (+/- 1 week) run-in period. The minimum and maximum values are 1-30, a lower score is regarded as more severe. Population: Full Analysis Set. A total of 230 subjects reported at least one intercourse attempt and had at least one IIEF assessment in a period for which at least one intercourse attempt was reported.
  score on a scale
    number analyzed (Participants) | 113 | 117 | 230
    (all) | 17.1 (5.9) | 17.1 (5.5) | 17.1 (5.7)

OUTCOME MEASURES:

1. Primary Outcome: Erectile Function (EF) Domain Score of the International Index of Erectile Function (IIEF)
Description: Erectile Function (EF) domain of the International Index of Erectile Function (IIEF) questionnaire. This will be measured at the end of the treatment periods of 4 weeks (+/- 1 week). The minimum and maximum values are 1-30, a lower score is regarded as more severe.
Time Frame: 4 Weeks
Population: Full Analysis Set. A total of 230 subjects reported at least one intercourse attempt and had at least one IIEF assessment in a period for which at least one intercourse attempt was reported. Observed cases only.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- MED Placebo: Participants who received MED Placebo. At least 4 applications of MED Placebo prior to intercourse in either the first or last 4 weeks of the study.
- MED2005: Participants who received MED2005 (0.2% glyceryl trinitrate gel). At least 4 applications of MED2005 prior to intercourse in either the first or last 4 weeks of the study.
Arm/Group | MED Placebo | MED2005
Number analyzed (Participants) | 225 | 223
score on a scale | 18.5 (6.7) | 19.6 (7.5)
Statistical Analysis 1: Comparison: MED Placebo vs MED2005; Test type: Superiority; p = 0.0132, Mixed Models Analysis; Mean Difference (Final Values) = 1.03, 95% CI 2-sided [0.22 to 1.84]

2. Secondary Outcome: Orgasmic Function Domain Score of the International Index of Erectile (IIEF)
Description: Orgasmic function domain of the International Index of Erectile Function (IIEF) questionnaire. This will be measured at the end of treatment periods of 4 weeks (+/- 1 week). The minimum and maximum values are 1-10, a lower score is regarded as having a worse outcome.
Time Frame: 4 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MED Placebo | MED2005
Number analyzed (Participants) | 225 | 223
score on a scale | 6.6 (2.6) | 7.0 (2.8)
Statistical Analysis 1: Comparison: MED Placebo vs MED2005; Test type: Superiority; p = 0.0122, Mixed Models Analysis; Mean Difference (Final Values) = 0.41, 95% CI 2-sided [0.09 to 0.73]

3. Secondary Outcome: Sexual Desire Domain Score of the International Index of Erectile Function (IIEF)
Description: Sexual desire domain of the International Index of Erectile Function (IIEF) questionnaire. This will be measured at the end of treatment periods of 4 weeks (+/- 1 week). The minimum and maximum values are 2-10, a lower score is regarded as having a worse outcome.
Time Frame: 4 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MED Placebo | MED2005
Number analyzed (Participants) | 225 | 222
score on a scale | 7.1 (1.8) | 7.5 (1.8)
Statistical Analysis 1: Comparison: MED Placebo vs MED2005; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.39, 95% CI 2-sided [0.21 to 0.57]

4. Secondary Outcome: Intercourse Satisfaction Domain Score of the International Index of Erectile Function (IIEF)
Description: Intercourse satisfaction domain of the International Index of Erectile Function (IIEF) questionnaire. This will be measured at the end of treatment periods of 4 weeks (+/- 1 week). The minimum and maximum values are 0-15, a lower score is regarded as having a worse outcome.
Time Frame: 4 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MED Placebo | MED2005
Number analyzed (Participants) | 223 | 223
score on a scale | 8.6 (2.8) | 9.0 (2.8)
Statistical Analysis 1: Comparison: MED Placebo; Test type: Superiority; p = 0.0055, Mixed Models Analysis; Mean Difference (Final Values) = 0.41, 95% CI 2-sided [0.12 to 0.69]

5. Secondary Outcome: Overall Satisfaction Domain Score of the International Index of Erectile Function (IIEF)
Description: Overall satisfaction domain of the International Index of Erectile Function (IIEF) questionnaire. This will be measured at the end of treatment periods of 4 weeks (+/- 1 week). The minimum and maximum values are 2-10, a lower score is regarded as having a worse outcome.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MED Placebo | MED2005
Number analyzed (Participants) | 225 | 222
score on a scale | 6.6 (2.2) | 7.1 (2.3)
Statistical Analysis 1: Comparison: MED Placebo vs MED2005; Test type: Superiority; p = 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.48, 95% CI 2-sided [0.20 to 0.76]

6. Secondary Outcome: Percentage of Affirmative Responses to Sexual Encounter Profile (SEP) Question 1
Description: SEP Question 1: "Were you able to achieve at least some erection (some enlargement of the penis)?". Answered yes/no after each intercourse event during treatment periods of 4 weeks (+/- 1 week). Assessed as a percentage of yes responses in each period.
Time Frame: 4 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of yes responses
Arm/Group | MED Placebo | MED2005
Number analyzed (Participants) | 225 | 228
percentage of yes responses | 86.93 (26.22) | 87.24 (26.47)
Statistical Analysis 1: Comparison: MED Placebo vs MED2005; Test type: Superiority; p = 0.7999, Generalized Linear Mixed Model; Means ratio = 0.995, 95% CI 2-sided [0.960 to 1.032]

7. Secondary Outcome: Percentage of Affirmative Responses to Sexual Encounter Profile (SEP) Question 2
Description: SEP Question 2: "Were you able to insert your penis into your partner's vagina?". Answered yes/no after each intercourse event during treatment periods of 4 weeks (+/- 1 week). Assessed as a percentage of yes responses in each period.
Time Frame: 4 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of yes responses
Arm/Group | MED Placebo | MED2005
Number analyzed (Participants) | 225 | 228
percentage of yes responses | 75.37 (34.91) | 75.53 (36.49)
Statistical Analysis 1: Comparison: MED Placebo vs MED2005; Test type: Superiority; p = 0.6746, Generalized Linear Mixed Model; Means ratio = 0.989, 95% CI 2-sided [0.937 to 1.043]

8. Secondary Outcome: Percentage of Affirmative Responses to Sexual Encounter Profile (SEP) Question 3
Description: SEP Question 3: "Did your erection last long enough for you to have successful intercourse?". Answered yes/no after each intercourse event during treatment periods of 4 weeks (+/- 1 week). Assessed as a percentage of yes responses in each period.
Time Frame: 4 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of yes responses
Arm/Group | MED Placebo | MED2005
Number analyzed (Participants) | 225 | 228
percentage of yes responses | 52.64 (38.81) | 57.32 (39.40)
Statistical Analysis 1: Comparison: MED Placebo vs MED2005; Test type: Superiority; p = 0.0959, Generalized Linear Mixed Model; Means ratio = 1.075, 95% CI 2-sided [0.987 to 1.170]

9. Secondary Outcome: Percentage of Affirmative Responses to Sexual Encounter Profile (SEP) Question 4
Description: SEP Question 4: "Were you satisfied with the hardness of your erection?". Answered yes/no after each intercourse event during treatment periods of 4 weeks (+/- 1 week). Assessed as a percentage of yes responses in each period.
Time Frame: 4 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of yes responses
Arm/Group | MED Placebo | MED2005
Number analyzed (Participants) | 225 | 228
percentage of yes responses | 28.97 (33.12) | 42.91 (41.0)
Statistical Analysis 1: Comparison: MED Placebo vs MED2005; Test type: Superiority; p < 0.0001, Generalized Linear Mixed Model; Means ratio = 1.522, 95% CI 2-sided [1.267 to 1.829]

10. Secondary Outcome: Percentage of Affirmative Responses to Sexual Encounter Profile (SEP) Question 5
Description: SEP Question 5: "Were you satisfied overall with this sexual experience?". Answered yes/no after each intercourse event during treatment periods of 4 weeks (+/- 1 week). Assessed as a percentage of yes responses in each period.
Time Frame: 4 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of yes responses
Arm/Group | MED Placebo | MED2005
Number analyzed (Participants) | 225 | 228
percentage of yes responses | 36.88 (36.98) | 48.23 (40.87)
Statistical Analysis 1: Comparison: MED Placebo vs MED2005; Test type: Superiority; p = 0.0005, Generalized Linear Mixed Model; Means ratio = 1.320, 95% CI 2-sided [1.128 to 1.545]

11. Secondary Outcome: Number of Participants With Affirmative Response to Global Assessment Questionnaire (GAQ) Question 1
Description: GAQ Question 1: "Has the treatment you have been taking improved your erectile function?". Answered yes/no after each treatment period of 4 weeks (+/- 1 week).
Time Frame: 4 Weeks
Population: Full Analysis Set. A total of 230 subjects reported at least one intercourse attempt and had at least one IIEF assessment in a period for which at least one intercourse attempt was reported. Complete cases only.
Measure: Count of Participants; unit: Participants
Arm/Group | MED Placebo | MED2005
Number analyzed (Participants) | 216 | 216
Participants | 56 | 94
Statistical Analysis 1: Comparison: MED Placebo vs MED2005; Test type: Superiority; p < 0.0001, Prescott Test (Exact)

12. Secondary Outcome: Number of Participants With Affirmative Response to Global Assessment Questionnaire (GAQ) Question 2
Description: GAQ Question 2: "Has the treatment improved your ability to engage in sexual activity?". Answered yes/no after each treatment period of 4 weeks (+/- 1 week).
Time Frame: 4 Weeks
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | MED Placebo | MED2005
Number analyzed (Participants) | 216 | 216
Participants | 54 | 85
Statistical Analysis 1: Comparison: MED Placebo vs MED2005; Test type: Superiority; p = 0.0003, Prescott Test (Exact)

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: Adverse events were assigned to a treatment as follows:
  * Period 1 treatment, if the onset date-time was on or after the first use of study medication of Period 1 and prior to the first study medication use of Period 2.
  * Period 2 treatment, if the onset date-time was on or after the first study medication use of Period 2.
  The number at risk are the number who actually used the corresponding treatment in the first and second intervention periods, subject to the cross-over sequence followed.
Arm/Group | MED Placebo | MED2005
All-Cause Mortality (participants affected / at risk) | 0/227 | 0/229
Serious Adverse Events (participants affected / at risk) | 0/227 | 0/229
Other Adverse Events (participants affected / at risk) | 15/227 | 28/229
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MED Placebo (N=227) | MED2005 (N=229)
Nasopharyngitis (Infections and infestations) | 11 | 13
Headache (Nervous system disorders) | 7 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other